CLINICAL TRIAL: NCT03244865
Title: Refinement of LaborView Electronic Fetal Monitor
Brief Title: Refinement of the OBMedical LaborView System
Status: Completed | Type: Observational
Sponsor: OBMedical Company (Other)
Collaborators: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: PRO00009835
Record Dates: First submitted 2017-08-03; First posted 2017-08-10 (Actual); Results first posted 2019-09-20 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-06

CONDITIONS: Fetal Monitoring

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Pregnant Females: All patients admitted to the Labor & Delivery Suite at UF Health, will be eligible for inclusion in the study except minors and those unable to consent for themselves.
  Nothing is required of the subjects. They will be non-invasively monitored for one to several hours. The information obtained will not be used for medical decision-making and there is no significant risk to the patient or her fetus. No longitudinal follow-up is planned or indicated.
  Interventions: Device: LaborView Electronic Fetal Monitor

INTERVENTIONS:
Device: LaborView Electronic Fetal Monitor — Per LaborView directions, electrode application sites will be prepared to reduce skin impedance, electrodes will be applied to the maternal abdomen and FHR data acquired for comparison with CTG data obtained through the traditional monitoring system. The comparison will be performed off-line.
  Nothing is required of the subjects. They will be non-invasively monitored for one to several hours. The information obtained will not be used for medical decision-making and there is no significant risk to the patient or her fetus.

SUMMARY:
Despite its limitations, fetal heart rate (FHR) tracing analysis is the best monitor of fetal well-being during labor or preparation for cesarean delivery. Current monitoring methods: transabdominal ultrasound (CTG: cardiotocograph) and fetal scalp electrodes (FSE) have limitations (tracing loss during fetal movement, potential to confuse maternal for fetal heart rate, inability to monitor during cesarean section or abdominal surgery) and, in the latter case, risks (infection, hematoma). A reliable, non-invasive monitor of the fetal heart rate that can be used during labor, non-obstetric and obstetric surgery during pregnancy is needed. Recent developments in use of maternal abdominal electrodes for extraction of the FHR and contraction information inform this study.

LaborView®, developed by researchers at University of Florida (UF) College of Medicine and OBMedical, is an FDA-approved non-invasive labor monitoring device. Refinement of the extraction algorithms continues, and that work is most effectively performed at UF, where the primary researchers and OBMedical are located.

LaborView monitoring will be recorded from up to150 subjects admitted to Labor and Delivery at UFHealth. Data will be simultaneously obtained from the standard labor monitor. These signals will then be analyzed off-line for comparison and refinement of algorithms.

DETAILED DESCRIPTION:
Despite its limitations, fetal heart rate (FHR) tracing analysis is the best monitor of fetal well being during labor. Typically, continuous electronic fetal monitoring is via transabdominal ultrasound (CTG: cardiotocograph). A transducer is strapped to the maternal abdomen and positioned in such a way to detect fetal rather than maternal heart rate. There are occasional periods of signal loss as the patient or her fetus moves, as well as times when the monitor incorrectly records the maternal signal. Maternal obesity presents particular challenges to non-invasive monitoring.

When there is particular concern regarding the fetal heart rate tracing the obstetrician may opt for a fetal scalp electrode (FSE). This is screwed into the fetus' presenting part through the opening in the cervix (requires ruptured membranes and adequate dilation). This signal is usually more reliable, but entails risks of chorioamnionitis, fetal scalp infection, scalp hematoma, and potential vertical transmission of maternal viruses including HIV and hepatitis.

Recently, devices have come to market that extract the FHR and uterine electromyograph (EMG) from maternal abdominal electrodes. The proposed study will provide data for refinement of the LaborView device produced by OBMedical.

Specific Aims:

The goal of this research is to evaluate the LaborView device under various settings and fetal heart rate accuracy as compared to a traditional CTG monitor.

Research Plan:

All patients admitted to the Labor & Delivery Suite at UF Health, will be eligible for inclusion in the study except minors and those unable to consent for themselves.

Following written informed consent, the external monitors (tocodynamometer and ultrasound) may not be removed. Per LaborView directions, electrode application sites will be prepared to reduce skin impedance, electrodes will be applied to the maternal abdomen and data acquired for comparison with CTG data obtained through the traditional monitoring system. FHR, ECG (electrocardiography), and uterine activity data from the existing fetal monitors will be collected via a laptop PC connected to the systems for comparison. The comparison will be performed off-line.

Evaluation of the data obtained will include (1) comparison of the calculated FHR with that of the CTG and/or fetal scalp electrode.

Nothing is required of the subjects. They will be non-invasively monitored for one to several hours. The information obtained will not be used for medical decision-making and there is no significant risk to the patient or her fetus. No longitudinal follow-up is planned or indicated.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to Labor and Delivery at Shands UF Health
* Are able to consent for themselves

Exclusion Criteria:

• Under the age of 18

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only Pregnant Females
Study Population: Pregnant Females admitted to Labor and Delivery at Shands UF Health who are over the age of 18 and able to consent themselves.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2016-09-29 (Actual); Primary Completion 2018-04-11 (Actual); Study Completion 2018-04-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida Shands Health, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Pregnant Females: All patients admitted to the Labor & Delivery Suite at UF Health, will be eligible for inclusion in the study except minors and those unable to consent for themselves.
  Nothing is required of the participants. They will be non-invasively monitored for one to several hours. The information obtained will not be used for medical decision-making and there is no significant risk to the patient or her fetus. No longitudinal follow-up is planned or indicated.
  LaborView Electronic Fetal Monitor: Per LaborView directions, electrode application sites will be prepared to reduce skin impedance, electrodes will be applied to the maternal abdomen and data acquired for comparison with CTG data obtained through the traditional monitoring system. FHR, ECG, and uterine activity data from the existing fetal monitors will be collected via a laptop PC connected to the systems for comparison. The comparison will be performed off-line.
Period: Overall Study
Arm/Group | Pregnant Females
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Pregnant Females: All patients admitted to the Labor & Delivery Suite at UF Health, will be eligible for inclusion in the study except minors and those unable to consent for themselves.
  Nothing is required of the subjects. They will be non-invasively monitored for one to several hours. The information obtained will not be used for medical decision-making and there is no significant risk to the patient or her fetus. No longitudinal follow-up is planned or indicated.
  LaborView Electronic Fetal Monitor: Per LaborView directions, electrode application sites will be prepared to reduce skin impedance, electrodes will be applied to the maternal abdomen and data acquired for comparison with CTG data obtained through the traditional monitoring system. FHR, ECG, and uterine activity data from the existing fetal monitors will be collected via a laptop PC connected to the systems for comparison. The comparison will be performed off-line.
Arm/Group | Pregnant Females
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27 (30.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 21
  More than one race | 2
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 35
Number of Subjects in active labor [Count of Participants; unit: Participants] | 35

OUTCOME MEASURES:

1. Primary Outcome: Fetal Heart Rate With the Laborview System Versus the CTG Monitor - Pilot Comparison Study
Description: Using standard of care CTG (Cardiotocography) already in place and the LaborView electrode-based FHR monitoring simultaneously, we will collect FHR data from both monitors simultaneously. We will compare the two FHR calculations using root mean squared error (RMSE).
Time Frame: 1 - 8 hours
Measure: Mean (90% Confidence Interval); unit: beats per minute
Groups:
- Pregnant Females: There is only one arm in this study. All monitored patients admitted to Labor & Delivery at UF Health, are eligible for inclusion in the study except minors and those unable to consent for themselves. They are non-invasively monitored for 1 to several hours. The information obtained is not used for medical decision-making and there is no significant risk to the patient or her fetus. No longitudinal follow-up is planned or indicated.
  All subjects in the study maintain the standard CTG monitoring they are using prior to enrollment in the study. The LaborView Electronic Fetal Monitor is added to the subject and both standard CTG FHR and LaborView FHR are collected simultaneously. LaborView electrode application sites are prepared to reduce skin impedance, and electrodes are applied to the maternal abdomen. The data collection laptop collects data from the standard monitor via serial port of the CTG and from LaborView via USB. The comparison of data is performed off-line.
Arm/Group | Pregnant Females
Number analyzed (Participants) | 35
beats per minute | 5.282 [4.8 to 5.75]
Statistical Analysis 1: Comparison: Pregnant Females; There is only one ARM in the study. Standard monitoring and LaborView monitoring will be collected simultaneously and analyzed; Test type: Non-Inferiority — Non-inferiority will be verified if the RMSE between the two systems is within 7 BPM. A complete power analysis was not included as this is a pilot study; p < .1, t-test, 2 sided — Pilot Study

ADVERSE EVENTS:
Time Frame: 11 months
Groups:
- Pregnant Females: All patients admitted to the Labor & Delivery Suite at UF Health, will be eligible for inclusion in the study except minors and those unable to consent for themselves.
  LaborView Electronic Fetal Monitor: Per LaborView directions, electrode application sites will be prepared to reduce skin impedance, electrodes will be applied to the maternal abdomen and data acquired for comparison with CTG data obtained through the traditional monitoring system. FHR, ECG, and uterine activity data from the existing fetal monitors will be collected via a laptop PC connected to the systems for comparison. The comparison will be performed off-line.
  Nothing is required of the participants. They will be non-invasively monitored for one to several hours. The information obtained will not be used for medical decision-making and there is no significant risk to the patient or her fetus.
Arm/Group | Pregnant Females
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2016-09-29): https://cdn.clinicaltrials.gov/large-docs/65/NCT03244865/Prot_000.pdf
  • Statistical Analysis Plan (2016-09-29): https://cdn.clinicaltrials.gov/large-docs/65/NCT03244865/SAP_001.pdf
  • Informed Consent Form (2016-09-29): https://cdn.clinicaltrials.gov/large-docs/65/NCT03244865/ICF_002.pdf